CLINICAL TRIAL: NCT02789423
Title: Clinical and Radiographical Evaluation of the Effect of Calcium Hydroxide Cement (Dycal) and Calcium Silicate Cement (Biodentine) in Direct Pulp Capping in Primary Teeth: a Randomized Clinical Trial
Brief Title: Clinical & Radiographical Evaluation of the Effect of Dycal & Biodentine in DPC in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modern Dental College and Research Centre, Indore (Other)
Responsible Party: Principal Investigator, Dr. Komal Gandhi, Post Graduate, Modern Dental College and Research Centre, Indore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ModernDCRC
Record Dates: First submitted 2016-04-13; First posted 2016-06-03 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Dental Pulp Exposure
MeSH Terms: conditions — Dental Pulp Exposure | interventions — tricalcium silicate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dycal (Active Comparator): Intervention: drug: Dycal, Other names: Calcium Hydroxide. Intervention Description:DPC using Dycal for direct pulp exposure was performed in 30 primary molar teeth after proper case selection.Clinical and radiographic evaluation was done.One month post operative criteria evaluated were-Clinical criteria:Spontaneous pain,Defective restoration/Recurrent caries,Sinus formation,TOP,Soft tissue swelling & Mobility. Radiographic criteria:Defective restoration/Recurrent caries,Periapical or furcal radiolucency,Pathological internal resorption,Replacement resorption,Intracanal calcification & Physiological resorption.The follow-up was at 3 and 6 months.
  Interventions: Procedure: Direct Pulp Capping using Dycal and Biodentine
- Biodentine (Active Comparator): Intervention: drug: Biodentine, Other names: Calcium Silicate. Intervention Description:DPC using Biodentine for direct pulp exposure was performed in 30 primary molar teeth after proper case selection.Clinical and radiographic evaluation was done.One month post operative criteria were-Clinical criteria:Spontaneous pain,Defective restoration/Recurrent caries,Sinus formation,TOP,Soft tissue swelling & Mobility.Radiographic criteria:Defective restoration/Recurrent caries, Periapical or furcal radiolucency,Pathological internal resorption,Replacement resorption,Intracanal calcification & Physiological resorption.The follow-up was at 3 and 6 months.
  Interventions: Procedure: Direct Pulp Capping using Dycal and Biodentine

INTERVENTIONS:
Procedure: Direct Pulp Capping using Dycal and Biodentine — The operative procedure performed as follows: i)Administration of L.A and rubber dam isolation. ii)High-speed carious enamel removal. iii)Dentine mechanical curettage. iv)Manual final dentine curettage using a spoon excavator. v)Hemorrhage control by cotton pellet moistened with 2.5% sodium hypochlorite placed over the exposure for 1-2min. vi)The exposure site would then be dried with sterile cotton pellet.The operator shall apply the pulp capping agent(dycal/Biodentine)according to the manufacturer's instructions.And then another cover of glass ionomer is applied.This would be followed by permanent restoration.
  Other Names: DPC

SUMMARY:
The purpose of this study was clinical and radiographical evaluation of the effect of calcium hydroxide cement (Dycal) and calcium silicate cement (Biodentine) in direct pulp capping in primary teeth.

DETAILED DESCRIPTION:
The aim of the present study is to compare Calcium Hydroxide cement (Dycal) ® and Calcium Silicate cement (Biodentine)TM as pulp capping agents in primary molars. The objective of this study include the evaluation of clinical and radiographic efficacy of Calcium Hydroxide cement (Dycal) ® and Calcium Silicate cement (Biodentine)TM, and their response in direct pulp capping treatment on primary molars during a 6 months follow up. After following the proper standardized procedure for direct pulp cap. In the current study direct pulp capping was performed using calcium hydroxide cement (Dycal)® and Calcium Silicate cement (Biodentine)TM on 60 primary teeth of children equally divided between 2 study groups randomly of both the sexes aged 4-9 years old. Complete case history was recorded in detail and intraoral periapical radiograph was also taken for teeth indicated for direct pulp capping. Written consent was obtained from the parents of participants before starting the procedure. Strict standardized procedure had been followed and the pulp capping agent (Dycal®/BiodentineTM) were applied according to the manufacturer's instructions.Each patient was evaluated clinically and radiographically for any abnormal clinical signs and symptoms at 1,3 and 6 months postoperatively.Better results for the success of the study could be relatively enhanced by close attention to rigid criteria for case selection, standardization of direct pulp capping procedure and meticulous performance of the procedure appear to be prerequisites for successful treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Good health.
2. Cooperative behaviour.
3. Informed consent from parents.
4. Primary molars with clinically active caries.
5. No history of spontaneous pain in teeth.
6. Restorable tooth with at least one half of root length present.
7. Absence of pathological mobility.
8. Absence of tenderness to percussion.
9. Normal gingiva and periodontal condition without the sign of pathology such as redness and swelling of vestibule, draining sinus tract or sensitivity to palpate in the vestibule.

In addition, the teeth treated by direct pulp capping had only a pin point mechanical exposure (0.5 to 1mm), for which haemorrhage control could be achieved within two minutes before proceeding with direct pulp capping.

Radiographically, there was absence of internal resorption, external resorption, periapical or furcation radiolucencies and pathology of succedenous permanent tooth follicle.

Exclusion Criteria:

* Patients with a history of spontaneous pain, tooth tender to percussion, absence of underlying permanent teeth, internal/external root resorption, apical/furcal lesions, sinus tract, physiologic or pathologic luxation, and/or presence of abscess were excluded from the study.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evidence of effectiveness of Dycal and Biodentine as Direct Pulp Capping agent in primary molars confirmed by clinical and radiographical evaluation. | 6 months
  Clinical Criteria: No spontaneous pain,Defective restoration/Recurrent caries,Sinus formation,TOP,Soft tissue swelling & Mobility. Radiographic criteria: No Defective restoration/Recurrent caries,Periapical or furcal radiolucency,Pathological internal resorption,Replacement resorption,Intracanal calcification & Physiological resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Komal IM Gandhi, BDS, Principal Investigator — DAVV; Dr. Mishthu Solanki, MDS, Study Chair — DAVV

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garrocho-Rangel A, Flores H, Silva-Herzog D, Hernandez-Sierra F, Mandeville P, Pozos-Guillen AJ. Efficacy of EMD versus calcium hydroxide in direct pulp capping of primary molars: a randomized controlled clinical trial. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 May;107(5):733-8. doi: 10.1016/j.tripleo.2008.12.017. Epub 2009 Feb 8. PMID 19201627
- [Background] Hilton TJ, Ferracane JL, Mancl L; Northwest Practice-based Research Collaborative in Evidence-based Dentistry (NWP). Comparison of CaOH with MTA for direct pulp capping: a PBRN randomized clinical trial. J Dent Res. 2013 Jul;92(7 Suppl):16S-22S. doi: 10.1177/0022034513484336. Epub 2013 May 20. PMID 23690353
- [Background] Fallahinejad Ghajari M, Asgharian Jeddi T, Iri S, Asgary S. Direct pulp-capping with calcium enriched mixture in primary molar teeth: a randomized clinical trial. Iran Endod J. 2010 Winter;5(1):27-30. Epub 2010 Feb 20. PMID 23130026
- [Background] Aminabadi NA, Farahani RM, Oskouei SG. Formocresol versus calcium hydroxide direct pulp capping of human primary molars: two year follow-up. J Clin Pediatr Dent. 2010 Summer;34(4):317-21. doi: 10.17796/jcpd.34.4.pntq604021604234. PMID 20831133
- [Background] Tuzuner T, Alacam A, Altunbas DA, Gokdogan FG, Gundogdu E. Clinical and radiographic outcomes of direct pulp capping therapy in primary molar teeth following haemostasis with various antiseptics: a randomised controlled trial. Eur J Paediatr Dent. 2012 Dec;13(4):289-92. PMID 23270285
- [Background] Shayegan A, Jurysta C, Atash R, Petein M, Abbeele AV. Biodentine used as a pulp-capping agent in primary pig teeth. Pediatr Dent. 2012 Nov-Dec;34(7):e202-8. PMID 23265156
- [Background] Asl Aminabadi N, Maljaei E, Erfanparast L, Ala Aghbali A, Hamishehkar H, Najafpour E. Simvastatin versus Calcium Hydroxide Direct Pulp Capping of Human Primary Molars: A Randomized Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2013 Winter;7(1):8-14. doi: 10.5681/joddd.2013.002. Epub 2013 Feb 21. PMID 23487477